CLINICAL TRIAL: NCT00742833
Title: A Randomized, Double Blind, Placebo Controlled, Phase II Study of KUC-7483 in Patients With Overactive Bladder
Brief Title: A Phase II Study of KUC-7483 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUC1203
Record Dates: First submitted 2008-08-05; First posted 2008-08-28 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Overactive Bladder (OAB)
Keywords: Overactive bladder; Frequency; Micturition; Urgency; Urge urinary incontinence; β3-agonist
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — ritobegron ethyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 (Experimental)
  Interventions: Drug: KUC-7483
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KUC-7483
  Arms: 3
Drug: Placebo
  Arms: 1

SUMMARY:
To investigate the efficacy and safety of KUC-7483 in overactive bladder patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptom of overactive bladder for more than 6 months.
* Patients who meet the following condition during the 3-day bladder diary period.

  * the mean number of micturitions per 24 hours is ≥8 times
  * the mean number of urgency episodes per 24 hours is ≥1 time

Exclusion Criteria:

* Patients who are diagnosed as stress urinary incontinence are predominant.
* Patients with urinary calculus, interstitial cystitis, or clinically significant urinary tract infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean number of micturitions per 24 hours | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in mean number of urgency episodes per 24 hours | 12 weeks
Change from baseline in mean number of incontinence episodes per 24 hours | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Omori, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (6):
- Japan (6):
  - Japan, Hokkaido Region
  - Japan, Kansai Region
  - Japan, Kanto Region
  - Japan, Kyushu Region
  - Japan, Shikoku Region
  - Japan, Tohoku Region